CLINICAL TRIAL: NCT01610037
Title: A Placebo and Active Controlled Study to Assess the Long-term Safety of Once Daily QVA149 for 52 Weeks in Chronic Obstructive Pulmonary Disease (COPD) Patients With Moderate to Severe Airflow Limitation
Brief Title: Comparison of Long-term Safety of the Combination Product QVA149A Against Placebo and Standard of Care Treatment in Chronic Obstructive Pulmonary Disease Patients With Moderate to Severe Airflow Limitation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQVA149A2339; 2012-002057-38 (EudraCT Number)
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: chronic obstructive pulmonary disease; COPD; QVA149; QAB149; NVA237; Indacaterol maleate; Glycopyronnium bromide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- QVA149 (Experimental)
  Interventions: Drug: QVA149
- Tiotropium (Active Comparator)
  Interventions: Drug: Tiotropium
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: QVA149 — QVA149 110/50 µg will be supplied as capsules in blister packs for once daily inhalation using the Novartis Concept1 SDDPI
  Arms: QVA149
Drug: Tiotropium — Tiotropium 18 µg will be supplied as capsules in blister packs for once daily inhalation using the HandiHaler SDDPI
  Arms: Tiotropium
Drug: placebo — placebo to QVA149A and Tiotropium will be supplied in the appropriate capsule in blister packs for use in either the Novartis Concept1 SDDPI or the HandiHaler SDDPI
  Arms: placebo

SUMMARY:
The study will assess the long-term safety of the fixed combination product QVA149 versus placebo and a standard of care treatment (tiotropium) in Chronic Obstructive Pulmonary Disease (COPD) patients with moderate to severe airflow limitation.

ELIGIBILITY:
Inclusion criteria:

* Male and female adults aged ≥40 years.
* Patients with stable COPD according to GOLD strategy (GOLD 2011).
* Patients with airflow limitation indicated by a post-bronchodilator FEV1 ≥ 30% and <80% of the predicted normal, and a post-bronchodilator.
* FEV1/FVC < 0.70.
* Current or ex-smokers who have a smoking history of at least 10 pack years.
* Patients with an mMRC ≥ grade 2

Exclusion criteria:

* History of long QT syndrome or prolonged QTc.
* Patients who have had a COPD exacerbation that required treatment with antibiotics and/or systemic corticosteroids and/or hospitalization in the 6 weeks prior to Visit 1.
* Patients with Type I or uncontrolled Type II diabetes.
* Patients with a history of asthma or have concomitant pulmonary disease.
* Patients with paroxysmal (e.g. intermittent) atrial fibrillation. Only patients with persistent atrial fibrillation and controlled with a rate control strategy for at least six months could be eligible.
* Patients who have clinically significant renal, cardiovascular, neurological, endocrine, immunological, psychiatric, gastrointestinal, hepatic, or hematological abnormalities which could interfere with the assessment of safety.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1215 (Actual)
Dates: Start 2012-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (95):
- Argentina (17):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Florida, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, San Isidro, Buenos Aires
  - Novartis Investigative Site, San Juan Bautista, Buenos Aires
  - Novartis Investigative Site, Vicente López, Buenos Aires
  - Novartis Investigative Site, Corrientes, Corrientes Province
  - Novartis Investigative Site, Concepción del Uruguay, Entre Ríos Province
  - Novartis Investigative Site, Mendoza, Mendoza Province
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
- Colombia (4):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Armenia
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
- Croatia (4):
  - Novartis Investigative Site, Sisak, Croatia
  - Novartis Investigative Site, Zagreb, Croatia
  - Novartis Investigative Site, Osijek
  - Novartis Investigative Site, Zagreb
- Estonia (2):
  - Novartis Investigative Site, Tartu, Estonia
  - Novartis Investigative Site, Tallinn
- Hungary (11):
  - Novartis Investigative Site, Cegléd, Hungary
  - Novartis Investigative Site, Debrecen, Hungary
  - Novartis Investigative Site, Érd, Hungary
  - Novartis Investigative Site, Monor, Hungary
  - Novartis Investigative Site, Siófok, Hungary
  - Novartis Investigative Site, Szarvas, Hungary
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Csorna
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Mosonmagyaróvár
- India (13):
  - Novartis Investigative Site, Hyderabad, A.p.
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Panjim, Goa
  - Novartis Investigative Site, Ahmedabad, India
  - Novartis Investigative Site, Nagpur - Maharashtra, India
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Trivandrum, Kerala
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Vellore, Tamil Nadu
- Israel (3):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
- Latvia (2):
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Mexico (3):
  - Novartis Investigative Site, León, Guanajuato
  - Novartis Investigative Site, Pachuca, Hidalgo
  - Novartis Investigative Site, Mexico City, Mexico City
- Novartis Investigative Site, Panama City, Provincia de Panamá, Panama
- Poland (4):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
- Russia (7):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Yaroslavl
- Serbia (2):
  - Novartis Investigative Site, Knez-Selo
  - Novartis Investigative Site, Kragujevac
- Novartis Investigative Site, Golnik, Slovenia
- South Korea (6):
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Pendik / Istanbul, Turkey
  - Novartis Investigative Site, Kartal
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Yenisehir/Izmir
- United Kingdom (10):
  - Novartis Investigative Site, Royal Leamington Spa, Warwickshire
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Cheshire
  - Novartis Investigative Site, Doncaster
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Merseyside
  - Novartis Investigative Site, Newport
  - Novartis Investigative Site, Portsmouth
  - Novartis Investigative Site, Wolverhampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2064 patients were screened, of whom 1216 patients were randomized to QVA149 110/50 µg o.d., tiotropium 18 µg o.d., or placebo. Of the 1216, one patient was randomized but not treated.
Pre-assignment Details: One patient of the 1216 was randomized but did not receive treatment
Groups:
- QVA149: 110/50 µg capsules for inhalation, o.d
- Tiotropium: 18 μg capsules for inhalation, o.d
- Placebo: To match QVA149 capsules for inhalation, o.d To match tiotropium capsules for inhalation, o.d
Period: All Patients
Arm/Group | QVA149 | Tiotropium | Placebo
Started | 407 | 405 | 404
Randomized Set (RAN) | 407 | 405 | 404
Full Analysis Set (FAS) | 407 | 405 | 403
Completed | 348 | 354 | 320
Not Completed | 59 | 51 | 84
Not completed — Adverse Event | 27 | 22 | 26
Not completed — Withdrawal by Subject | 12 | 10 | 20
Not completed — Unsatisfactory therapeutic effect | 9 | 8 | 27
Not completed — Death | 4 | 2 | 1
Not completed — Protocol deviation | 4 | 3 | 3
Not completed — Abnormal laboratory value | 1 | 1 | 0
Not completed — Administrative problems | 1 | 4 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Abnormal test procedure result(s) | 0 | 1 | 3
Period: Treatment and Follow up Period
Arm/Group | QVA149 | Tiotropium | Placebo
Started | 407 | 405 | 404
Completed | 382 | 377 | 378
Not Completed | 25 | 28 | 26
Not completed — Subject withdrew consent | 13 | 14 | 16
Not completed — Death | 10 | 5 | 4
Not completed — Administrative problems | 1 | 3 | 2
Not completed — Lost to Follow-up | 1 | 6 | 4

BASELINE CHARACTERISTICS:
Population: The RAN included all randomized patients regardless of whether or not they actually received study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | QVA149 | Tiotropium | Placebo | Total
Number analyzed (Participants) | 407 | 405 | 404 | 1216
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (7.89) | 64.1 (8.57) | 64.9 (7.95) | 64.5 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 105 | 94 | 318
  Male | 288 | 300 | 310 | 898

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Serious Adverse Events
Description: The overall rate of serious adverse events reported from initiation through 30 days post last dose.
Time Frame: Week 52
Population: The safety set included all patients who received at least one dose of study drug and had at least one post-baseline safety assessment. Patients were analyzed according to treatment received. A patient who had no adverse events also constitutes a safety assessment.
Measure: Number; unit: Participants
Groups:
- Tiotropium 18 µg o.d: 18 μg capsules for inhalation, o.d
Arm/Group | QVA149 | Tiotropium 18 µg o.d | Placebo
Number analyzed (Participants) | 407 | 403 | 402
Participants | 55 | 55 | 50

2. Secondary Outcome: Percentage of Patients With Composite Endpoint of All-cause Mortality, and Serious Cardio- and Cerebrovascular (CCV) Events.
Description: The endpoint of all-cause mortality and serious CCV events (composite) was chosen to further characterize any discernible risks. The patients with an event in the analysis were those who had at least one of the 2 events namely, all-cause mortality and serious CCV, during treatment or within 30 days after the date of last dose of study drug.
Time Frame: 52 weeks
Population: The full analysis set (FAS) included all randomized patients who received at least one dose of study drug. Patients were analyzed according to the treatment they were assigned to at randomization. If the patient was assigned to the wrong stratum for randomization, the patient was analyzed according to the actual (rather than assigned) stratum.
Measure: Number; unit: Percentage of participants
Arm/Group | QVA149 | Tiotropium 18 µg o.d | Placebo
Number analyzed (Participants) | 407 | 405 | 403
Percentage of participants | 3.9 | 2 | 1

3. Secondary Outcome: Post-hoc Analysis: Percentage of Patients With Composite Endpoint of Cardiovascular Death and MACE
Description: The composite endpoint included all deaths and all serious CCV events, including MACE and events which were not considered MACE. A rigorous post hoc analysis was done on composite endpoint of CV deaths and major adverse cardiovascular events (MACE). The patients with an event in the analysis were those who had at least one of the 2 events namely, CV deaths and MACE, during treatment or within 30 days after the date of last dose of study drug.
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | QVA149 | Tiotropium 18 µg o.d | Placebo
Number analyzed (Participants) | 407 | 405 | 403
Percentage of participants | 1 | 0.7 | 0.7

4. Secondary Outcome: Change From Baseline in Pre-Dose Forced Expiratory Volume Over in Second (FEV1)
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. Baseline FEV1 was defined as the average of the pre-dose FEV1 measured at -45 minutes (min) and -15 min at day 1.
Time Frame: Day 22, 43, 85, 183, 274 and 364
Population: The full analysis set (FAS) included all randomized patients who eceived at least one dose of study drug. Patients were analyzed according to the treatment they were assigned to at randomization. If the patient was assigned to the wrong stratum for randomization, the patient was analyzed according to the actual (rather than assigned) stratum
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Tiotropium 18 µg o.d | Placebo
Number analyzed (Participants) | 407 | 405 | 379
Liters
  Day 22 (n=378, 383, 361) | 0.1733 (0.18537) | 0.1018 (0.18389) | -0.0148 (0.16758)
  Day 43 (n=380, 375, 345) | 0.1751 (0.20800) | 0.0961 (0.18261) | -0.0196 (0.18178)
  Day 85 (n=373, 373, 340) | 0.1752 (0.20198) | 0.0785 (0.19606) | -0.0506 (0.19369)
  Day 183 (n=356, 358, 314) | 0.1557 (0.21754) | 0.0714 (0.20358) | -0.0583 (0.20305)
  Day 274 (n=343, 351, 303) | 0.1463 (0.21424) | 0.0750 (0.21489) | -0.0601 (0.20936)
  Day 364 (n=333, 346, 297) | 0.1468 (0.22933) | 0.0559 (0.22433) | -0.0826 (0.21443)

5. Secondary Outcome: Change From Baseline in Health Status as Measured by St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C)
Description: The SGRQ-C contains 40 items divided into two parts covering three aspects of health related to COPD: Part I covers "Symptoms" and is concerned with respiratory symptoms, their frequency and severity; Part II covers "Activity" and is concerned with activities that cause or are limited by breathlessness; Part II is also concerned with "Impacts" which covers a range of aspects concerned with social functioning and psychological disturbances resulting from airways disease. A score will be calculated for each of these three subscales and a "Total" score will also be calculated. In each case the lowest possible value is zero and the highest 100. Higher values correspond to greater impairment of health status.
Time Frame: Measurment at day 364
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | QVA149 | Tiotropium 18 µg o.d | Placebo
Number analyzed (Participants) | 343 | 349 | 314
Score | -6.79 (12.611) | -6.12 (13.695) | -2.18 (13.311)

6. Secondary Outcome: Change From Baseline in Daily, Morning and Evening Symptom Scores
Description: Patients will be provided with an electronic diary (eDiary) to record daily clinical symptoms, or rescue medication. The patients will be instructed to routinely complete the patient diary twice daily. There are 9 total symptom questions for a total possible score of 27 at each timepoint. A higher score means the patient is reporting more symptoms related to Chronic Obstructive Pulmonary Disease. The mean daily total symptom score, the mean daytime total symptom score and the mean nighttime total symptom score were calculated for each patient over 52 weeks. Diary data recorded during the 14 day run-in period were used to calculate the baseline.
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | QVA149 | Tiotropium 18 µg o.d | Placebo
Number analyzed (Participants) | 407 | 405 | 403
Score
  Daily total symptom score (n=395, 395, 385) | -1.3478 (1.91692) | -1.2283 (1.93241) | -0.7683 (1.73598)
  Daytime total symptom score (n= 380, 385, 374) | -1.1688 (1.93350) | -1.0669 (1.90366) | -0.5641 (1.62577)
  Nighttime total symptom score (n= 387, 388, 375) | -0.9731 (1.96898) | -0.9532 (1.78168) | -0.5984 (1.73356)

7. Secondary Outcome: Change From Baseline in Percentage of Nights With 'no Nighttime Awakenings
Description: A night with 'no nighttime awakenings' is defined from diary data as any night where the patient did not wake up due to symptoms.
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of nights
Arm/Group | QVA149 | Tiotropium 18 µg o.d | Placebo
Number analyzed (Participants) | 387 | 388 | 375
Percentage of nights | 11.34 (30.115) | 10.66 (26.579) | 8.21 (28.002)

8. Secondary Outcome: Change From Baseline in Percentage of no Daytime Symptoms
Description: A day with 'no daytime symptoms' is defined from the diary data as any day where the patient has recorded in the evening no cough, no wheeze, no production of sputum and no feeling of breathlessness (other than when running) during the past 12 hours (approx. 8 am to 8 pm).
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | QVA149 | Tiotropium 18 µg o.d | Placebo
Number analyzed (Participants) | 380 | 385 | 374
Percentage of days | 5.56 (19.670) | 4.72 (15.942) | 1.78 (15.733)

9. Secondary Outcome: Change From Baseline in Percentage of Days Able to Perform Usual Daily Activities.
Description: A day able to perform usual daily activities' is defined from diary data as any day where the patient was not prevented from performing their usual daily activities due to respiratory symptoms.
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | QVA149 | Tiotropium 18 µg o.d | Placebo
Number analyzed (Participants) | 380 | 385 | 374
Percentage of days | 10.79 (31.006) | 6.54 (30.215) | 1.13 (25.039)

10. Secondary Outcome: Change From Baseline in 1 Hour Post-dose Forced Vital Capacity (FVC) Measurements
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards
Time Frame: Day 1, 22, 43, 85, 183, 274 and 364
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QVA149 | Tiotropium 18 µg o.d | Placebo
Number analyzed (Participants) | 407 | 405 | 403
Liters
  Day 1(n=403, 402, 399) | 0.3331 (0.30312) | 0.2806 (0.28293) | 0.0630 (0.22884)
  Day 22 (n=384, 381, 362) | 0.3971 (0.40009) | 0.3123 (0.36755) | 0.0178 (0.33624)
  Day 43 (n=380, 373, 351) | 0.4021 (0.42797) | 0.2966 (0.37124) | 0.0274 (0.35681)
  Day 85 (376, 371, 345) | 0.4169 (0.42175) | 0.2867 (0.40131) | 0.0035 (0.36897)
  Day 183 (n=364, 359, 317) | 0.3880 (0.45342) | 0.2822 (0.39781) | -0.0283 (0.36919)
  Day 274 (n=349, 352, 306) | 0.3582 (0.43072) | 0.2821 (0.40546) | -0.0404 (0.37777)
  Day 364 (n= 336, 347, 302) | 0.3153 (0.46560) | 0.2224 (0.40778) | -0.0498 (0.39908)

11. Secondary Outcome: Time to Premature Discontinuation
Description: Time to premature treatment discontinuation for each treatment group was displayed using a Kaplan-Meier curve. The date of last dose of study medication was considered as the event date and also as the censoring date for those patients who did not discontinue treatment early. The range of the 'time to treatment discontinuation' varied from 5-407 days in the Tiotropium group. Hence the model estimated lower limit of the median time to treatment discontinuation is greater than the scheduled treatment period of 52 weeks.
Time Frame: Time varied from 5 - 407 days
Population: The Safety set consisted of all patients that received at least one dose of study medication and had at least one post-baseline safety assessment. Patients were analyzed according to treatment received.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | QVA149 | Tiotropium 18 µg o.d | Placebo
Number analyzed (Participants) | 407 | 405 | 403
Days | NA [NA to NA] — NA - insufficient number of participants with events | NA [378 to NA] — NA - insufficient number of participants with events | NA [NA to NA] — NA - insufficient number of participants with events

12. Secondary Outcome: Change From Baseline in 1 Hour Post-dose FEV1 Measurements
Description: The avg 60 min post dose forced expiratory volume in 1 second (FEV1) at visit 4, 5, 6, 7, 8 and 9 will be analyzed.
Time Frame: Day 1, 22, 43, 85, 183, 274 and 364
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QVA149 | Tiotropium 18 µg o.d | Placebo
Number analyzed (Participants) | 407 | 405 | 403
Liters
  Day 1 (n=403, 402, 399) | 0.2064 (0.14248) | 0.1567 (0.13349) | 0.0281 (0.11123)
  Day 22 (n=384, 381, 362) | 0.2883 (0.21074) | 0.2077 (0.20027) | 1.5827 (15.69990)
  Day 43 (n=380, 373, 351) | 0.2904 (0.23377) | 0.2008 (0.20752) | 1.6209 (16.89209)
  Day 85 (n=376, 371, 345) | 0.3026 (0.23260) | 0.1913 (0.23274) | -0.0217 (0.20195)
  Day 183 (n=364, 359, 317) | 0.2860 (0.24351) | 0.1842 (0.22851) | -0.0253 (0.21129)
  Day 274 (n=349, 352, 306) | 0.2749 (0.24314) | 0.1681 (0.23626) | -0.0360 (0.21854)
  Day 364 (n= 336, 347, 302) | 0.2619 (0.25967) | 0.1621 (0.23922) | -0.0533 (0.21560)

ADVERSE EVENTS:
Groups:
- QVA 149: 110/50 µg capsules for inhalation, o.d
Arm/Group | QVA 149 | Tiotropium | Placebo
Serious Adverse Events (participants affected / at risk) | 55/407 | 55/405 | 50/403
Other Adverse Events (participants affected / at risk) | 294/407 | 294/405 | 309/403
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA 149 (N=407) | Tiotropium (N=405) | Placebo (N=403)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 3 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 2 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Hypothermia (General disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Pneumonia (Infections and infestations) | 3 | 6 | 2
Pneumonia bacterial (Infections and infestations) | 2 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Arteriogram coronary (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1 | 0
Radiculitis (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
VIth nerve paresis (Nervous system disorders) | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 20 | 18 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 1
Ischaemia (Vascular disorders) | 0 | 0 | 1
Jugular vein distension (Vascular disorders) | 1 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA 149 (N=407) | Tiotropium (N=405) | Placebo (N=403)
Influenza (Infections and infestations) | 7 | 11 | 18
Lower respiratory tract infection (Infections and infestations) | 22 | 14 | 19
Nasopharyngitis (Infections and infestations) | 33 | 31 | 26
Respiratory tract infection viral (Infections and infestations) | 4 | 11 | 7
Upper respiratory tract infection (Infections and infestations) | 18 | 22 | 18
Upper respiratory tract infection bacterial (Infections and infestations) | 27 | 28 | 25
Viral upper respiratory tract infection (Infections and infestations) | 19 | 13 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 6 | 6
Headache (Nervous system disorders) | 9 | 13 | 11
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 269 | 274 | 287
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 21 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 12
Hypertension (Vascular disorders) | 9 | 10 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.